CLINICAL TRIAL: NCT00544297
Title: A Multi-center, Open-label Study to Examine the Safety and Toleration of 0.05% PEP005 Topical Gel in Patients With Actinic Keratoses on the Dorsum of the Hand
Brief Title: A Study to Examine the Safety and Toleration of PEP005 Topical Gel in Patients With Actinic Keratoses on the Top of the Hand
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Collaborators: Omnicare Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-018
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Topical; Dermatology; Hand
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEP005 gel administration (Experimental): 0.05% PEP005 Topical Gel administered for two consecutive days to a 25cm2 contiguous AK treatment area on the top of the hand
  Interventions: Drug: PEP005 gel

INTERVENTIONS:
Drug: PEP005 gel — Two day application, 0.05%
  Other Names: PEP005

SUMMARY:
The purpose of this study is to examine the safety and toleration of PEP005 Topical Gel, administered on an actinic keratosis (AK) treatment area on the top of a hand.

DETAILED DESCRIPTION:
Actinic keratoses (AK) is a common skin condition characterized by rough, scaly patches or sores on the top layer of the skin which if left untreated can progress to skin cancer. Current treatments can cause scarring and hypopigmentation, be inconvenient, or require long treatment duration. Non-invasive alternative therapy for treatment of AK lesions is thus being researched.

ELIGIBILITY:
Inclusion Criteria:

* Male patients at least 18 years of age.
* Post-menopausal female patients
* 4 to 8 clinically typical, visible and discrete AK lesions within an area on the dorsum of one hand.
* Written informed consent has been obtained.
* Agreement from the patient to allow photographs of the selected AK treatment area to be taken and used as part of the study data package.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs); and Local Skin Responses (LSR) | 57 days

SECONDARY OUTCOMES:
The complete clearance rate of AK lesions; partial clearance rate of AK lesions and baseline clearance rate of AK lesions. | 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Arthur P Bertolino, MD, Study Director — Chief Medical Officer and VP Medical Affairs
Locations (4):
- United States (4):
  - Skin Surgery Medical Group Inc, San Diego, California
  - Gwinnett Clinical Research Centre, Snellville, Georgia
  - Dermatology Clinical Research Centre of San Antonio, San Antonio, Texas
  - Dermatology Associates of Tyler, Tyler, Texas

REFERENCES:
- See also: Food and Drug Administration — http://www.fda.gov/
- See also: Human Research Ethics Committee — http://www.quorumreview.com